CLINICAL TRIAL: NCT05313048
Title: The APSantiCo Observational Study - Prospective Observational Study to Evaluate a Possible Change in APS Antibody Profiles After COVID-19 Infection or Vaccination
Brief Title: Prospective Observational Study to Evaluate a Possible Change in APS Antibody Profiles After COVID-19 Infection or Vaccination
Acronym: APSantiCo
Status: Completed | Type: Observational
Sponsor: Cardioangiologisches Centrum Bethanien (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. E. Lindhoff-Last, Clinical Professor, Cardioangiologisches Centrum Bethanien
Other Study IDs: APSantiCo-Study
Record Dates: First submitted 2022-04-05; First posted 2022-04-06 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Antiphospholipid Syndrome; COVID-19 Infection; COVID-19 Vaccination
MeSH Terms: conditions — Antiphospholipid Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — frozen citrated plasma samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study to evaluate a possible change in APS antibody profiles after COVID-19 infection or vaccination

DETAILED DESCRIPTION:
Prospective observational study to evaluate a possible change in antiphospholipid antibody profiles after coronavirus disease 2019 (COVID-19) infection or vaccination.

Patients with antiphospholipid syndrome (APS) with thromboembolic complications recorded using the retrospective database of the APSANTICO registry (ClinicalTrials.gov Identifier: NCT05195372) will serve as a baseline for a prospective observational study to investigate the extent to which COVID 19 infection and/or COVID 19 vaccination alters APS antibody profiles.

Current literature suggests that patients who have been or are infected with COVID-19 are at higher risk of thrombosis. This increased risk is due to, among other things, damaged endothelium, slower blood flow and observed hypercoagulability of the blood.

It has also been described that COVID-19 patients may have a higher prevalence of lupus anticoagulant. Based on these assumptions, one of the aims of the prospective observational study is to determine whether and to what extent COVID-19 infection affects the antibody profile of APS patients.

In addition, atypical thrombosis with thrombocytopenia has been repeatedly reported recently as a rare side effect after COVID-19 vaccination with two recombinant adenoviral vectors encoding the spike protein antigen of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) (ChAdOx1 nCov-19, AstraZeneca and Ad26.COV2.S, Johnson&Johnson).

The extent to which thrombosis could also occur after messenger RNA (mRNA) vaccines has not yet been clearly proven.

Furthermore, it is unclear whether COVID-19 infections and/or vaccinations can possibly influence the expression and level of antiphospholipid antibody titres. Therefore, another aim of the prospective observational study is to compare the antiphospholipid antibody results available from the retrospective registry before COVID-19 vaccination or COVID-19 infection with the antibody results after COVID-19 infection and/or vaccination. For this purpose, the patients who were recorded in the retrospective register are contacted by post with an information letter and then called in by telephone to the investigators coagulation centre for a follow-up examination after the COVID-19 vaccinations have been carried out and/or after COVID-19 infection. Then, during this examination, a blood sample is taken to monitor the course of the antiphospholipid antibodies. In addition, patients are offered a test of COVID-19 nucleocapsid antibodies and COVID-19 spike antibodies free of charge to check the success of the vaccination. This is of particular interest as some of these patients are taking immunosuppressive drugs due to an underlying autoimmune disease, which could weaken the immune response.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Confirmed antiphospholipid syndrome with thromboembolic clinical manifestations (venous thromboembolism, pulmonary embolism, thrombophlebitis etc.)
* Patients with APS antibody risk profile (single/double/triple positivity)
* Written consent for participation in the prospective APSantiCo observational study

Exclusion Criteria:

* APS with isolated pregnancy complications
* No anticoagulation medication
* Inadequately diagnosed APS
* Non-compliance on the part of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with antiphospholipid syndrome with thromboembolic clinical manifestations (venous thromboembolism, pulmonary embolism, thrombophlebitis etc.) or Patients with APS antibody risk profile (single/double/triple positivity)
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
change in APS antibody status after surviving COVID-19 infection and/or receiving COVID-19 vaccination | 2015-2022
  The main observational variable is the change in APS antibody status in patients with antiphospholipid syndrome after surviving COVID-19 infection and/or receiving COVID-19 vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Edelgard Lindhoff-Last, Prof. MD, Study Chair — Cardioangiology Center Bethanien
Locations (1):
- Cardioangiology Center Bethanien (CCB), Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: No